CLINICAL TRIAL: NCT03642262
Title: A Phase I, Open-label, Single Dose, Randomized, 2-way Crossover Bioequivalence Study Comparing Mucinex® Extended Release 600 mg Bi-Layer Tablet to a Reference Immediate Release Guaifenesin Tablet (Taken as 200 mg Every 4 Hours [q4h] x 3 Doses) in Normal Healthy Volunteers
Brief Title: Mucinex® ER 600 mg Bi-layer Tablet Versus Guaifenesin Immediate Release (IR) 200 mg q4h
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Inc. (Industry)
Responsible Party: Sponsor
Organization: Reckitt Benckiser LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-MUC-02
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Acetylcysteine; Guaifenesin

STUDY DESIGN:
Intervention Model Description: 2-Way Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A: Mucinex® ER 600 mg (Experimental): Mucinex® ER 600 mg bi-layer single dose tablet by mouth under fasting condition.
  Interventions: Drug: Mucinex®
- Treatment B: Guaifenesin 200 mg (Active Comparator): Guaifenesin 200 mg immediate release (IR) tablet thrice (at 0, 4, and 8 hours) by mouth under fasting condition.
  Interventions: Drug: Mucinex®

INTERVENTIONS:
Drug: Mucinex® — Mucinex® 600 mg single dose ER bi-layer tablet
  Other Names: guaifenesin

SUMMARY:
Demonstrate bioequivalence of guaifenesin in Mucinex® extended release (ER) 600 mg tablet in normal healthy volunteers compared to the immediate release guaifenesin 200 mg tablet reference product marketed

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been obtained (i.e. be informed of the nature of the study and give written consent prior to any study procedure). Able to read, understand, and sign the informed consent, after the nature of the study has been explained.
2. Age: 18 to 55 years of age, inclusive.
3. Sex: Male or female.
4. Status: Healthy subjects.
5. BMI: ≥18.0 and ≤28.0 kg/m2.
6. No clinically significant findings in vital signs measurements at screening.
7. No clinically significant abnormal laboratory values at screening.
8. No clinically significant findings from a 12-lead electrocardiogram (ECG) at screening.
9. Have no significant diseases or clinically relevant medical condition in the opinion of the investigator.
10. Males who participate in this study are willing to:

    * remain abstinent [not engage in sexual intercourse] from the start of drug administration until 90 days after the end of the study or
    * use (or their partner will use, as applicable) two effective methods of birth control [condom, diaphragm, cervical cap, vaginal sponge, spermicide, IUD, tubal ligation, vasectomy, or hormonal contraceptives] from the start of drug administration until 90 days after the end of the study.

    Females who participate in this study are:
    * unable to have children (e.g., post-menopausal, hysterectomy);
    * willing to remain abstinent [not engage in sexual intercourse] from 21 days prior to drug administration until 30 days after the end of the study; or
    * willing to use two effective methods of birth control [condom, diaphragm, cervical cap, vaginal sponge, spermicide, non-hormonal Intrauterine Device (IUD) (in place for 3 months), tubal ligation, partner has vasectomy, hormonal contraceptives for 3 months prior to drug administration] from 30 days prior to drug administration until 30 days after the end of the study.
11. Have no clinically significant findings from a physical examination.

Exclusion Criteria:

Subjects to whom any of the following conditions apply must be excluded:

1. Employee of Pharma Medica Research Inc. (PMRI) or Reckitt Benckiser.
2. Partner or first-degree relative of any Investigator at PMRI.
3. Known history or presence of any clinically significant medical condition.
4. Known or suspected carcinoma.
5. Presence of hepatic or renal dysfunction.
6. Presence of clinically significant gastrointestinal disease or history of malabsorption within the last year.
7. Known history or presence of galactose or fructose intolerance, sucrase-isomaltase insufficiency, Lapp lactase insufficiency, galactosemia, or glucose-galactose malabsorption syndrome.
8. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
9. History of drug or alcohol or medicinal product addiction requiring treatment within the past two years or excessive alcohol consumption (more than 10 units per week) Note: one unit is defined as 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of spirits
10. Positive test result for serum Human Chorionic Gonadotropin (hCG) consistent with pregnancy (females only), HIV, Hepatitis B surface antigen or Hepatitis C antibody.
11. Positive test result for urine drugs of abuse (cannabinoids, opiates, amphetamines, cocaine, phencyclidine, tricyclic antidepressants, barbiturates, methadone and benzodiazepines) or urine cotinine.
12. Difficulty fasting or consuming standard meals.
13. Females who are lactating.
14. Does not tolerate venipuncture.
15. Use of tobacco or nicotine-containing products within 12 months prior to drug administration.
16. On a special diet within 30 days prior to drug administration (e.g., liquid, protein, raw, food diet).
17. Donation or loss of whole blood (including clinical trials):

    * ≥50 ml and ≤499 ml within 30 days prior to drug administration
    * ≥500 ml within 56 days prior to drug administration.
18. Females who have started taking hormonal contraceptives or have changed their method or brand of hormonal birth control within 3 months prior to drug administration.
19. Have had a tattoo or body piercing within 30 days prior to drug administration.
20. Use of drugs of the monoamine oxidase inhibitor (MAOI) class within 30 days prior to drug administration.
21. Known history or presence of hypersensitivity, intolerance or idiosyncratic reaction to guaifenesin or any other drug substances with similar activity.
22. Previously enrolled in this study.
23. Participated in another clinical trial or received an investigational product within 30 days prior to drug administration.
24. Unable in the opinion of the Investigator to comply fully with the study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06-02 (Actual); Primary Completion 2013-08-09 (Actual); Study Completion 2013-08-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre study conducted in Canada.
Pre-assignment Details: Total Thirty (30) subjects were enrolled in the study among them 27 subjects completed the study.
Groups:
- Cohort 1 (Mucinex First Then Guaifenesin): Treatment A : Mucinex® ER 600 mg bi-layer single dose tablet by mouth under fasting condition.
  Treatment B : Guaifenesin 200 mg immediate release (IR) tablet q4h (total of 3 doses) by mouth under fasting condition.
  Cohort 1
  Period 1 - Treatment A or Treatment B at Sequence AB.
  Period 2 - Treatment B or Treatment A at Sequence BA.
  Scheduled Washout of 7 days between drug administrations.
- Cohort 2 (Guaifenesin Then Mucinex): Treatment A : Mucinex® ER 600 mg bi-layer single dose tablet by mouth under fasting condition.
  Treatment B : Guaifenesin 200 mg immediate release (IR) tablet q4h (total of 3 doses) by mouth under fasting condition.
  Cohort 2
  Period 1 - Treatment A or Treatment B at Sequence AB.
  Period 2 - Treatment B or Treatment A at Sequence BA.
  Scheduled Washout of 7 days between drug administrations.
Period: Period 1
Arm/Group | Cohort 1 (Mucinex First Then Guaifenesin) | Cohort 2 (Guaifenesin Then Mucinex)
Started | 12 | 18
Completed | 11 | 16
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout: 7 Days
Arm/Group | Cohort 1 (Mucinex First Then Guaifenesin) | Cohort 2 (Guaifenesin Then Mucinex)
Started | 11 | 16
Completed | 11 | 16
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Cohort 1 (Mucinex First Then Guaifenesin) | Cohort 2 (Guaifenesin Then Mucinex)
Started | 11 | 16
Completed | 11 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Treatment A : Mucinex® ER 600 mg bi-layer single dose tablet by mouth under fasting condition.
  Treatment B : Guaifenesin 200 mg immediate release (IR) tablet q4h (total of 3 doses) by mouth under fasting condition.
  Cohort 1
  Period 1 - Treatment A or Treatment B at Sequence AB.
  Period 2 - Treatment B or Treatment A at Sequence BA.
  Scheduled Washout of 7 days between drug administrations.
  Cohort 2
  Period 1 - Treatment A or Treatment B at Sequence AB.
  Period 2 - Treatment B or Treatment A at Sequence BA.
  Scheduled Washout of 7 days between drug administrations.
Arm/Group | Overall Study
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Age Group [Count of Participants; unit: Participants]
  18 to 40 years | 14
  41 to 64 years | 16
Height [Mean (Standard Deviation); unit: cm] | 167.4 (9.1)
Weight [Mean (Standard Deviation); unit: kg] | 67.2 (9.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 23.9 (2.2)
Race [Number; unit: participants]
  Asian | 5
  Black or African American | 6
  White | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Guaifenesin
Description: Maximum measured analyte concentration over the sampling period.
Time Frame: 0 (pre-dose) ,0.25,0.5, 0.75, 1,1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14, 16, 20 and 24 hours
Population: Pharmacokinetic (PK) Parameter Set Population includes all subjects from the PK dataset with evaluable PK parameters for each treatment period.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Test: RB Mucinex® ER 600 mg: Mucinex® ER 600 mg bi-layer single dose tablet by mouth under fasting condition.
- Reference: Guaifenesin 200 mg: Guaifenesin 200 mg immediate release (IR) tablet q4h (total of 3 doses) by mouth under fasting condition.
Arm/Group | Test: RB Mucinex® ER 600 mg | Reference: Guaifenesin 200 mg
Number analyzed (Participants) | 27 | 27
ng/ml | 1076.37 (414.80) | 1223.89 (522.04)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUCt) of Guaifenesin
Description: The area under the analyte concentration versus time curve, from time zero (0) to the time of the last measurable analyte concentration (t), as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Population: PK Dataset
Measure: Mean (Standard Deviation); unit: ng·h/ml
Arm/Group | Test: RB Mucinex® ER 600 mg | Reference: Guaifenesin 200 mg
Number analyzed (Participants) | 27 | 27
ng·h/ml | 4288.30 (1654.57) | 4641.48 (2211.99)

3. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Guaifenesin
Description: Time of the maximum measured analyte concentration over the sampling period.
Time Frame: as for outcome 1
Population: PK Dataset
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Test: RB Mucinex® ER 600 mg | Reference: Guaifenesin 200 mg
Number analyzed (Participants) | 27 | 27
hr | 0.75 (0.33) | 1.45 (2.43)

4. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time 0 to Infinity (AUCinf) of Guaifenesin
Description: AUCinf = AUCt + Cp/Kel, where Cp is the predicted analyte concentration at the time of the last measurable analyte concentration.
Time Frame: as for outcome 1
Population: PK Dataset
Measure: Mean (Standard Deviation); unit: ng·h/ml
Arm/Group | Test: RB Mucinex® ER 600 mg | Reference: Guaifenesin 200 mg
Number analyzed (Participants) | 27 | 27
ng·h/ml | 4306.21 (1658.06) | 4647.47 (2212.37)

5. Secondary Outcome: Terminal Elimination Rate Constant (Kel) of Guaifenesin
Description: Elimination rate constant calculated from the slope of the terminal portion of the plasma profile calculated by least squares regression of log (concentration) versus time
Time Frame: as for outcome 1
Population: PK Dataset
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Test: RB Mucinex® ER 600 mg | Reference: Guaifenesin 200 mg
Number analyzed (Participants) | 27 | 27
1/h | 0.4727 (0.1711) | 0.7635 (0.1011)

6. Secondary Outcome: Terminal Elimination Half-life (T½) of Guaifenesin
Description: Terminal elimination half-life, calculated from the equation: T½ = In(2)/Kel.
Time Frame: as for outcome 1
Population: PK Dataset
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Test: RB Mucinex® ER 600 mg | Reference: Guaifenesin 200 mg
Number analyzed (Participants) | 27 | 27
h | 1.70 (0.75) | 0.93 (0.15)

7. Secondary Outcome: Relative Bioavailability (RF) of Guaifenesin
Description: RF is measured by (AUCinf ER / AUCinf IR) x (ER dose / IR dose)
Time Frame: as for outcome 1
Population: Outcome involved analyzing data from both intervention groups (ER and IR) in combination as per the provided formula, therefore, separate analysis for each intervention cannot be reported
Measure: Mean (Standard Deviation); unit: ng·h/ml
Groups:
- All Study Participants: Mucinex® ER 600 mg bi-layer single dose tablet by mouth under fasting condition.
  Guaifenesin 200 mg immediate release (IR) tablet q4h (total of 3 doses) by mouth under fasting condition.
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
ng·h/ml | 0.9542 (0.1770)

8. Secondary Outcome: Number of Adverse Events(AEs) Experienced by Participants
Description: Intensity determination Mild=AE does not limit usual activities; subject may experience slight discomfort Moderate=AE results in some limitation of usual activities;subject may experience significant discomfort Severe=AE results in an inability to carry out usual activities; subject may experience intolerable discomfort or pain Unassessable/Unclassifiable=Insufficient information to be able to make an assessment Conditional/Unclassified=Insufficient information to make an assessment at present (causality is conditional on additional information) Unrelated=No possibility that the AE was caused by study drug Unlikely=Slight, but remote, chance that the AE was caused by study drug, but the balance of judgment is that it was most likely not due to the study drug Possible=Reasonable suspicion that the AE was caused by the study drug Probable=Most likely that the AE was caused by study drug Certain=The AE was definitely caused by study drug Investigational Medicinal Product (IMP)
Time Frame: Up to period 2 (8.3 days/200 hours)
Population: Safety population
Measure: Number; unit: Events
Arm/Group | Test: RB Mucinex® ER 600 mg | Reference: Guaifenesin 200 mg
Number analyzed (Participants) | 28 | 29
Events
  TEAE by severity: Mild | 1 | 9
  TEAE by severity: Moderate | 0 | 0
  TEAE by severity: Severe | 0 | 0
  Relationship to IMP: Unassessable/Unclassifiable | 0 | 3
  Relationship to IMP: Conditional /Unclassified | 0 | 0
  Relationship to IMP: Unrelated | 0 | 0
  Relationship to IMP: Unlikely | 0 | 0
  Relationship to IMP: Possible | 1 | 6
  Relationship to IMP: Probable | 0 | 0
  Relationship to IMP: Certain | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 8.3 days (200 hours)
Groups:
- Treatment B: Guaifenesin 200 mg: Guaifenesin 200 mg immediate release (IR) tablet q4h (total of 3 doses) by mouth under fasting condition.
Arm/Group | Treatment A: Mucinex® ER 600 mg | Treatment B: Guaifenesin 200 mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 1/28 | 4/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Mucinex® ER 600 mg (N=28) | Treatment B: Guaifenesin 200 mg (N=29)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 1 (1)
Catheter site swelling (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No